CLINICAL TRIAL: NCT00558584
Title: Multicentre, Randomized, Double-blind, Prospective Investigation on the Effects of Immunoadsorption on Cardiac Function in Patients With Dilated Cardiomyopathy
Brief Title: Multicenter Study of Immunoadsorption in Dilated Cardiomyopathy
Acronym: IASO-DCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Krupp von Bohlen und Halbach-Foundation, Essen, Germany (Unknown); ENDI-Foundation, Bad Homburg, Germany (Unknown); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA-2006-001
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dilated Cardiomyopathy
Keywords: dilated cardiomyopathy; immunoadsorption; immunoglobulin G
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IA/IgG group (Active Comparator): immunoadsorption using IA columns and subsequent IgG substitution
  Interventions: Device: protein A immunoadsorption
- control group (Placebo Comparator): pseudo-immunoadsorption followed by an intravenous infusion without IgG
  Interventions: Device: pseudo-immunoadsorption

INTERVENTIONS:
Device: protein A immunoadsorption — protein-A immunoadsorption and i.v. IgG substitution
  Arms: IA/IgG group
Device: pseudo-immunoadsorption — pseudo-immunoadsorption followed by an intravenous infusion without IgG
  Arms: control group

SUMMARY:
The purpose of this study is to investigate the effects of immunoadsorption and subsequent IgG substitution in patients with dilated cardiomyopathy compared to a control group.

DETAILED DESCRIPTION:
Dilated cardiomyopathy (DCM) is characterized by ventricular chamber enlargement and systolic dysfunction with normal LV wall thickness. According to reports heretofore, the incidence of this disorder in industrialized Western countries lies within the order of magnitude of 5 - 8 new illnesses per year for every 100,000 population. The prevalence, accordingly, is approximately 36 patients for every 100,000 population. However, recent data suggest higher actual prevalence of DCM: at present the estimated prevalence of congestive heart failure ranges from 2% to 6%. According to recently published studies (e.g., the MERIT-HF study and the COPERNICUS study), about 30% to 35% of patients with congestive heart failure suffer from non-ischemic myocardial heart disease. DCM was diagnosed, furthermore, in 12% of the patients of the CIBIS II study. Approximately 26% of the patients with reduced left-ventricular systolic function from the CHARM-added study suffered from heart failure due to DCM. Based on these data, assumption is justified that in Germany approximately 500,000 patients suffer from DCM. Despite advances in medical treatment of heart failure, the general prognosis for DCM is poor. In many cases, treatment options are surgical e.g., heart transplantation or implantation of an assist device.

An association between virus myocarditis and DCM has been hypothesized for a subset of patients with DCM. Both experimental and clinical data indicate that viral infection and inflammatory processes are involved in the pathogenesis of myocarditis and DCM, and may represent important factors causing progression of ventricular dysfunction.

Abnormalities of the cellular immune system are present in patients with myocarditis and DCM. For patients with DCM, immunohistological methods have been introduced for diagnosis of myocardial inflammation. Infiltration with lymphocytes and mononuclear cells as well as increased expression of cell adhesion molecules, are frequent phenomena in DCM. These findings support the hypothesis that the immune process is still active. Furthermore, activation of the humoral immune system with production of cardiac antibodies plays an important role in DCM. Several antibodies against cardiac structures have been detected in DCM patients - including antibodies that act against mitochondrial proteins, alpha- and beta-cardiac myosin heavy chain isoforms, the cardiac beta-receptor, the muscarinic acetylcholine receptor-2, and the sarcolemmal Na-K-ATPase. The functional significance of cardiac autoantibodies is under debate. It is possible that autoantibodies are formed as a consequence of inflammatory reactions to cellular destruction, in which case they should be regarded as an epiphenomenon. Cardiac autoantibodies, on the other hand, may likewise play an active role in the pathogenesis of DCM by triggering the disease process, or by contributing to development of myocardial contractile dysfunction. For certain antibodies, in-vitro data indicate a negative effect on cardiac performance. In myocarditis and DCM, heart-reactive cytotoxic auto-antibodies to the ADP/ATP carrier were found. These antibodies cross-react with the calcium channel of the cardiomyocytes. Purified antibodies obtained from DCM patients induce a negative inotropic effect in isolated rat cardiomyocytes by decreasing the calcium transients. Immunization of rodents against peptides derived from cardiovascular G-protein receptors induces morphological changes of myocardial tissue resembling DCM. Furthermore, recent data have provided evidence those antibodies against the beat1-receptor itself induce DCM: rats immunized against the second extracellular loop of cardiac beta1-receptors develop progressive left ventricular dilatation and dysfunction. Interestingly, sera transferred from these immunized animals to unsensitized rats induced the similar cardiomyopathic phenotype, thus demonstrating the pathogenic potential of a particular antibody for development of DCM. Further confirmation of the principle that autoantibodies contribute to induction of the disease process and to progression to DCM has been provided in a recent study. The authors showed that mice deficient in the programmed cell death-1 (PD-1) immunoinhibitory co-receptor develop autoimmune DCM with production of high-titre circulating IgG autoantibodies reactive to a 33-kilodalton protein expressed specifically on the surface of cardiomyocytes. This antigen was recently identified as cardiac troponin I.

When cardiac antibodies impair cardiac function, their removal would logically be expected to lead to an improvement in the patient's haemodynamic situation. Cardiac antibodies belong to the IgG fraction and can be eliminated by immunoadsorption (IA) therapy. Immunoadsorption has been introduced as a method for treatment of autoimmune processes e.g., Goodpasture's syndrome and lupus erythematodes. This form of therapy has already been successfully applied for treatment of DCM. Several pilot studies have shown that IA improves cardiac function in patients with DCM. The first uncontrolled pilot study disclosed acute beneficial haemodynamic effects of IA in patients with severe heart failure due to DCM. A randomized study followed, to investigate the haemodynamic effects of additional IA therapy for DCM. This study included patients with DCM (NYHA III-IV, LVEF <30%) who were under stable medication. In the IA group, IA was conducted on three consecutive days, with one IA session daily. On the grounds of safety - i.e., to reduce the risk of infection after immunoglobulin depletion - immunoglobulin G was substituted after the last IA session. Immunoadsorption and subsequent IgG substitution (IA/IgG) was repeated for 3 courses at monthly intervals until month 3. In contrast to the control group, patients in the IA/IgG group demonstrated after 3 months a significant increase in cardiac index (CI), paralleled by a similar increase in stroke volume index. A recent study demonstrated that IA/IgG therapy likewise mitigates the inflammatory process in the myocardium of DCM patients. A case-controlled study, performed by others, conducted IA in one course of 5 consecutive days without IgG substitution subsequent to immunoglobulin depletion. This study did not repeat IA during follow-up. In this study, LVEF increased from 22 to 40% one year after IA: a significant gain in contrast to the control group without IA therapy.

Recent data indicate that the beneficial haemodynamic effects of IA are related to removal of negative inotropic cardiac antibodies. Detection of cardio-depressant antibodies in the plasma of DCM patients, before IA, effectively predicts acute and prolonged haemodynamic improvement during IA. A further study clearly disclosed that the cardio depressant antibodies belong to the IG-3 subclass [38]. The removal of antibodies of the IgG-3 subclass accordingly represents an essential mechanism in IA therapy of DCM.

Protein-A and anti-IgG columns are licensed for IA. Anti-IgG sepharose effectively eliminates all IgG subclasses, including IgG-3. Protein A binds to the Fc part of human IgG-1, -2, -4. However, the affinity of protein A to IgG-3 is low. IgG-3 removal can be markedly increased by protein-A, through the use of an optimized treatment regime, by prolonging the IA course to 4 - 5 sessions, and by reducing the loading volume of the protein columns with plasma. In use of this adsorption regime for IgG-3 elimination, protein-A IA induces significant acute and prolonged haemodynamic improvement of DCM patients. Furthermore, IA treatment with protein A adsorption performed in 1 course on 5 consecutive days induces improvement of the left ventricular function of DCM patients over a period of 6 months, with results comparable to those received by IA treatment repeated in 4 courses at monthly intervals. Despite optimized medical treatment, the prognosis of DCM is still poor. For most patients, heart transplantation will represent the only palliative treatment option. Alternative therapeutic strategies for treatment of DCM are consequently of essential interest.

This randomized multicentre study will investigate for the first time by means of a double-blind study design whether a specific causal intervention - i.e., the removal of autoantibodies - will influence the disease process and improve the cardiac function of patients suffering from heart failure due to DCM.

ELIGIBILITY:
Inclusion Criteria:

* Dilated cardiomyopathy
* LVEF <= 40% determined by contrast echocardiography
* NYHA class II - IV
* Age 18 - 70
* Disease duration: symptomatic heart failure ≥ 6 months and <7 years prior to screening date
* Treatment with ACE inhibitors or angiotensin II receptor blockers (ARB), beta-blockers, and aldosterone antagonists (the latter at the discretion of the attending physician), for at least 6 months and at stable doses for at least 2 months prior to screening date.
* The patient's informed consent

Exclusion Criteria:

* NYHA class IV patients who are bed-ridden and dependent upon parenteral medication
* Cardiac insufficiency resulting from another basic disease (e.g. coronary artery disease, ≥50% stenosis of major vessel as ascertained by coronary angiography performed more recent than three years before screening date, hypertensive heart disease, or valvular defects >second degree
* History of myocardial infarction
* Acute myocarditis according to Dallas criteria
* Endocrine disorder excluding insulin-dependent diabetes mellitus
* Implanted cardiac defibrillator (ICD) <1 month before screening date
* Cardiac resynchronization therapy (CRT) <6 months before screening date
* I.v. medication with inotropic drugs, vasodilators or repeated (>1/day) i.v. administration of diuretics.
* Active infectious disease, or signs of ongoing infection with CRP >10mmol/L
* Impaired renal function (serum creatinine >220 µmol/L)
* Any disease requiring immunosuppressive drugs
* Anaemia (haemoglobin below 90 g/L) due to other causes than CHF
* Pregnancy or lactation, or childbearing potential without appropriate contraception
* Alcohol or drug abuse
* Presence of a malignant tumour, or remission of malignancy < 5 years
* Refusal of the patient to provide consent
* Suspected poor capability to follow instructions and cooperate
* Another life-threatening disease with poor prognosis (survival less than 2 years)
* Participation in any other clinical study within less than 30 days prior to screening date
* Previous treatments with IA or immunoglobulin
* Contraindications for application of the echocardiography contrast agent used (in accordance to the product specification). [Amendment 8]

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-12; Primary Completion 2021-09 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) at rest, as determined by contrast echocardiography | six months

SECONDARY OUTCOMES:
Clinical outcome (non-cardiovascular death, cardiovascular death, sudden death, hospitalization for cardiovascular cause/heart failure, acute myocardial infarction, unstable angina, stroke, cardiac interventions/procedures, clinical deterioration) | 24 months
LVEF at rest, as determined by contrast echocardiography | 12 and 24 months
Reduction of brain natriuretic peptides (BNP and/or NT pro-BNP) | 6, 12, and 24 months
Cardiopulmonary exercise capacity | 6, 12, and 24 months
LVEF at rest, as determined by magnetic resonance imaging (optional) | 6, 12, and 24 months
Serious clinical adverse events | day 7, 1 month, and 6 months
Quality of life (MLHFQ) | 6, 12, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephan B Felix, MD, Principal Investigator — Ernst-Moritz-Arndt University
Locations (21):
- Germany (19):
  - Deutsches Herzzentrum München, München, Bavaria
  - Medizinische Klinik und Poliklinik I (Campus Großhadern u. Campus Innenstadt), München, Bavaria
  - Kerckhoff-Klinik Forschungsgesellschaft mbH, Bad Nauheim
  - Herz- und Diabeteszentrum NRW, Klinik für Thorax- und Kardiovaskularchirurgie, Bad Oeynhausen
  - Herz- und Diabeteszentrums NRW, Bad Oeynhausen
  - Medizinische Klinik und Poliklinik, Kardiologie, Angiologie, Pneumologie , Charité, Universitätsmedizin Berlin, Campus Mitte, Berlin
  - Kardiologie (CC11), Campus Virchow, Charité, Universitätsmedizin Berlin, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Medizinische Klinik und Poliklinik II, Universitätsklinkum Bonn, Bonn
  - Klinik für Kardiologie, Westdeutsches Herzzentrum Essen, Universität Duisburg-Essen, Essen
  - Abteilung Kardiologie und Pneumologie, Universität Göttingen - Bereich Humanmedizin, Göttingen
  - Klinik für Innere Medizin B, Universität Greifswald, Greifswald
  - Klinik für Innere Medizin III, Medizinische Universitätsklinik Heidelberg, Heidelberg
  - Kardiologie, Angiologie und Internistische Intensivmedizin, Universitätsklinik Homburg/Saar, Homburg (Saar)
  - Klinik für Innere Medizin I, Universitätsklinikum Jena, Jena
  - Universitätsklinikum Magdeburg, Universitätsklinik für Kardiologie, Magdeburg
  - Abteilung Kardiologie und Pulmologie, Robert-Bosch-Krankenhaus, Stuttgart
  - Medizinische Klinik und Poliklinik, Abteilung Innere Medizin III, Medizinische Univ.-Klinik Tübingen, Tübingen
  - Medizinische Klinik und Poliklinik I, Klinikum der Bayrischen Julius-Maximilians-Universität, Würzburg
- Internal Medicine - Cardiology, Belgrade University School of Medicine, Belgrade, Serbia
- Department of Cardiology, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Staudt A, Staudt Y, Dorr M, Bohm M, Knebel F, Hummel A, Wunderle L, Tiburcy M, Wernecke KD, Baumann G, Felix SB. Potential role of humoral immunity in cardiac dysfunction of patients suffering from dilated cardiomyopathy. J Am Coll Cardiol. 2004 Aug 18;44(4):829-36. doi: 10.1016/j.jacc.2004.04.055. PMID 15312867
- [Background] Felix SB, Staudt A, Landsberger M, Grosse Y, Stangl V, Spielhagen T, Wallukat G, Wernecke KD, Baumann G, Stangl K. Removal of cardiodepressant antibodies in dilated cardiomyopathy by immunoadsorption. J Am Coll Cardiol. 2002 Feb 20;39(4):646-52. doi: 10.1016/s0735-1097(01)01794-6. PMID 11849864
- [Background] Staudt A, Schaper F, Stangl V, Plagemann A, Bohm M, Merkel K, Wallukat G, Wernecke KD, Stangl K, Baumann G, Felix SB. Immunohistological changes in dilated cardiomyopathy induced by immunoadsorption therapy and subsequent immunoglobulin substitution. Circulation. 2001 Jun 5;103(22):2681-6. doi: 10.1161/01.cir.103.22.2681. PMID 11390337
- [Background] Staudt A, Bohm M, Knebel F, Grosse Y, Bischoff C, Hummel A, Dahm JB, Borges A, Jochmann N, Wernecke KD, Wallukat G, Baumann G, Felix SB. Potential role of autoantibodies belonging to the immunoglobulin G-3 subclass in cardiac dysfunction among patients with dilated cardiomyopathy. Circulation. 2002 Nov 5;106(19):2448-53. doi: 10.1161/01.cir.0000036746.49449.64. PMID 12417541
- [Background] Felix SB, Staudt A. Non-specific immunoadsorption in patients with dilated cardiomyopathy: mechanisms and clinical effects. Int J Cardiol. 2006 Sep 10;112(1):30-3. doi: 10.1016/j.ijcard.2006.05.014. Epub 2006 Jul 21. PMID 16860418
- See also: Homepage: Department of Internal Medicine B, Ernst-Moritz-Arndt University, Greifswald, Germany — http://www.medizin.uni-greifswald.de/inn_b/